CLINICAL TRIAL: NCT04836585
Title: Technology-Enabled (Electronic) Measurement Based Care(MBC) for Perinatal Depression and Anxiety: A Pilot Randomized Controlled Trial
Brief Title: eMBC for Perinatal Depression and Anxiety
Acronym: eMBC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Women's College Hospital (Other)
Responsible Party: Principal Investigator, Simone Vigod, Chief, Department of Psychiatry, Women's College Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 2020-0090-B
Record Dates: First submitted 2021-03-31; First posted 2021-04-08 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Depression, Postpartum; Anxiety
Keywords: Measurement based care
MeSH Terms: conditions — Depression, Postpartum; Anxiety Disorders

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: The RA randomizing the participant will be not be blinded to the treatment allocation because they have to inform the provider of the treatment allocation. This RA will not be collecting outcome measures. The RA collecting outcome measures will be blinded to the treatment allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Care As Usual (No Intervention): Participants in the control condition are followed by their RLS psychiatrists during the study as per usual care.
- eMBC Intervention (Experimental): Participants in the intervention arm are followed by their RLS psychiatrists during the study at clinically appropriate intervals with the addition of eMBC.
  Interventions: Other: eMBC Intervention

INTERVENTIONS:
Other: eMBC Intervention — The treating psychiatrist sets a flag in the patient's electronic chart that prompts them to complete self-report scales prior to each appointment:
  1. Edinburgh Postnatal Depression Scale (EPDS) for symptoms of depression and anxiety
  2. PROMIS Neuro-QOL and PROMIS ASCQ-Me Social Functioning Short form for measures of functional capacity
  3. Adapted Frequency, Intensity, and Burden Side Effects Rating (FIBSER) Scale for participants taking antidepressant medication to measure side effects
  Patient participants and providers can view the questionnaire results over time in the electronic chart item by item, and/or see them in graphical format. During the clinical encounter, the provider and patient participant review the results of the scales, as part of a collaborative re-evaluation of the treatment plan.
  Arms: eMBC Intervention

SUMMARY:
Depression and anxiety that occur around the time of pregnancy can adversely impact a person's health and well-being, and their child's health and development. Fewer than 20% of affected people are adequately treated, often because of under-use of medications. Measurement based care (MBC) is a model of care where psychiatric symptoms are routinely tracked and reviewed together by a patient and their doctor to better manage symptoms. It has not been systematically evaluated for perinatal depression and anxiety. The overall objective of this study is to test the feasibility of MBC in this population to inform a future large randomized controlled trial for definitive evaluation. In order to avoid known barriers to MBC, electronic MBC (eMBC) will be used. With eMBC, patients can enter their symptoms into their electronic medical records before their appointment so that they can be evaluated by their doctor during the appointment. In this pilot study, the feasibility of recruitment for a future efficacy trial, including feasibility of recruitment, and retention, acceptability and adherence to a trial protocol will be evaluated.

DETAILED DESCRIPTION:
A parallel group randomized controlled trial (RCT) will be conducted. Eligible and consenting patients with depression and/or anxiety will be randomized in a 1:1 ratio to either the eMBC condition or a control condition. The study will be stratified by diagnosis (major depressive disorder vs generalized anxiety disorder).

80 patient participants will be recruited from the Reproductive Life Stages (RLS) Program at Women's College Hospital. The active treatment phase of the study is 12 weeks.

Outcomes will be measured online and by phone at 4-, 8-, and 12- weeks post-randomization. Following the completion of the study, some participants will be asked to participate in follow-up interviews. RLS psychiatrists whose patients participated in the study will participate in a focus group.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18
2. Currently pregnant or mother* of a live infant 0-12 months of age and living at the same residence

   *Through natural birth, adoption, surrogacy, including cis women, non-binary and transgender people in all their diversity
3. EPDS >12 at enrollment

Exclusion Criteria:

1. Active suicidal ideation, substance abuse or dependence
2. Current or past mania or psychosis or current major depressive episode with psychosis

4. Incapable of consenting to participation 5. Unable to read or unable to speak English

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2022-01-04 (Actual); Primary Completion 2023-10-27 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Feasibility of the trial protocol: Recruitment | 12 weeks post randomization
  Measures of recruitment include rate of recruitment and reason for non-participation.
Feasibility of the trial protocol: Participant Acceptability | 12 weeks post randomization
  Surveys and interviews will be used to capture data relating to perceived usefulness and acceptability of technology and its perceived benefit. These will be combined to capture an overall acceptability measure.
Feasibility of the trial protocol: Provider Acceptability | 12 weeks post randomization
  Surveys and focus groups will be used to capture data relating to usability and tolerability of eMBC in clinical practice.
Feasibility of the trial protocol: Adherence | 12 weeks post randomization
  Chart review will be used to measure the number of visits, the proportion of visits with completed scales and which scales were completed, proportion of visits where review of symptom scales was documented in the patient record, the proportion of visits where providers recorded that they used the data from symptom scales to inform the treatment, and proportion of visits where medication was started, changed, dose adjusted or stopped. These will be combined to provide an overall measure of how closely the intervention protocol was followed.

SECONDARY OUTCOMES:
Clinical outcomes - clinician-assessed depression symptoms | 4, 8, and 12 weeks post randomization
  The Montgomery-Asberg Depressive Rating Scale (MADRS) is a standard clinician-administered measure of depressive symptoms with good reliability and validity in clinical populations. The MADRS has good responsiveness to the effect of anti-depressant treatments. The 17-items are rated on a 7-point (0-6) (score range 0-60), with lower scores indicating fewer symptoms of depression and higher scores indicating a higher degree of symptoms.
Clinical outcomes - self-report depression symptoms | each clinical appointment up to 12 weeks post randomization
  Depressive symptoms will be measured using the Edinburgh Postnatal Depressive Scale (EPDS), a self-report scale that has been validated for use in pregnancy and postpartum. EPDS scores range from 0 to 30. EPDS scores >12 are predictive of a diagnosis of depression, with higher scores indicating more severe symptoms.
Clinical outcomes - anxiety symptoms | 4, 8, and 12 weeks post randomization
  The Hamilton Anxiety Rating Scale (HAM-A) is a clinician-rated measure that assesses the severity of symptoms of anxiety. The HAM-A has good reliability and validity in populations with depression and anxiety. The 14-items are rated on a 5-point scale (0-4) with scores ranging from 0-56. Scores <17 indicate mild severity, 18-24 mild to moderate severity and 25-30 moderate to severe symptoms.
Clinical outcomes - functional capacity | each clinical appointment up to 12 weeks post randomization
  The PROMIS Neuro-QOL - Ability to Participate in Social Roles and Activities - Short Form is a brief self-report tool used to measure functional capacity.
Clinical outcomes - social functioning | each clinical appointment up to 12 weeks post randomization
  PROMIS ASCQ-Me Social Functioning - Short Form is a brief self-report tool used to measure functional capacity.
Clinical outcomes - antidepressant side effects | each clinical appointment up to 12 weeks post randomization
  The Frequency, Intensity, and Burden Side Effects Rating (FIBSER) Scale is a brief 3-item scale used to measure three domains of anti-depressant side effects including frequency, intensity, and burden of antidepressant medication. The last question relating to burden is scored 0-6 with low scores indicating no medication adjustment is needed, and high scores indicating that the dose needs to be decreased or the medication changed.

OTHER OUTCOMES:
Co-variates: Participants | Baseline
  Sociodemographic, obstetrical, and psychiatric history data will be collected on the Baseline Questionnaire. A diagnostic phone interview using the Mini International Neuropsychiatric Interview (MINI) will be conducted for major depressive disorder, obsessive-compulsive disorder, panic disorder, agoraphobia, social anxiety disorder, generalized anxiety disorder and post-traumatic stress disorder.
Co-variates: Providers | Baseline
  Provider co-variates including age, number of years in practice, familiarity with technology, use of technology in their practice, and use of MBC prior to this study.

CONTACTS AND LOCATIONS:
Overall Officials: Renu Gupta, MD, Principal Investigator — Women's College Hospital
Locations (1):
- Women's College Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Askari N, Gupta R, Hussain-Shamsy N, Barker LC, Champagne T, Lam RW, Bishop K, Pirmohamed J, Michalowska M, Shah V, Katzman H, Jalan A, Shanmuganathan A, Wang V, Vigod SN. Electronic Measurement-based care (eMBC) for perinatal depression and anxiety: a pilot randomized controlled trial. BMC Psychiatry. 2025 Apr 29;25(1):437. doi: 10.1186/s12888-025-06876-3. PMID 40301831